CLINICAL TRIAL: NCT01661686
Title: A Randomized Comparison of a Fully Covered Self Expandable Metal Stent Versus a Partially Covered Self Expandable Metal Stent in Malignant Esophageal Strictures
Brief Title: Fully Covered or Partially Covered Stents in Malignant Esophageal Strictures
Acronym: COPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Principal Investigator, Manon Spaander, M.D., PhD, Foundation for Liver Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPAC
Record Dates: First submitted 2012-08-01; First posted 2012-08-09 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Esophageal Cancer; Esophageal Stenosis
Keywords: esophageal cancer; esophageal stenosis; stent; endoscopy
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insertion of a partially covered SEMS (Active Comparator)
  Interventions: Device: Partially covered SEMS
- Insertion of a Fully covered SEMS (Active Comparator)
  Interventions: Device: Fully covered SEMS

INTERVENTIONS:
Device: Partially covered SEMS — Boston Scientific, Natick, United States diameter 18 mm, lengths of 10, 12 and 15 cm available
  Other Names: WallFlex Partially covered esophageal stent
  Arms: Insertion of a partially covered SEMS
Device: Fully covered SEMS — Boston Scientific, Natick, United States diameter 18 mm, lengths of 10, 12 and 15 cm available
  Other Names: WallFlex Fully covered esophageal stent
  Arms: Insertion of a Fully covered SEMS

SUMMARY:
The purpose of this study is to determine whether fully covered or partially covered metal stents are more favorable in incurable malignant stenosis of the esophagus or cardia. Primary outcome will be the occurence of recurrent dysphagia which is defined as dysphagia due to a stent or tumour related cause in a 6-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Malignant stricture of the esophagus or cardia
* No curative treatment options available
* Dysphagia grade of at least 2 (i.e. swallow semi-solid foods or less)
* Informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Previous treatment with self-expandable metal stent for same condition
* Evidence of tumor within 2 cm of the upper esophageal sphincter.
* Presence of an esophago-tracheal or -bronchial fistula or both.
* Not able to undergo upper endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco J Bruno, M.D., Prof, Study Director — Erasmus Medical Center
Locations (5):
- Netherlands (5):
  - IJsselland Hospital, Capelle aan den IJssel, South Holland
  - Sint Fransiscus Gasthuis, Rotterdam, South Holland
  - Ikazia Hospital, Rotterdam, South Holland
  - Albert Schweitzer Hospital, Zwijndrecht, South Holland
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Derived] Didden P, Reijm AN, Erler NS, Wolters LMM, Tang TJ, Ter Borg PCJ, Leeuwenburgh I, Bruno MJ, Spaander MCW. Fully vs. partially covered selfexpandable metal stent for palliation of malignant esophageal strictures: a randomized trial (the COPAC study). Endoscopy. 2018 Oct;50(10):961-971. doi: 10.1055/a-0620-8135. Epub 2018 Jun 12. PMID 29895072

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS
Started | 49 | 49
Completed | 47 | 47
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — did not receive allocated intervention | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient, which was allocated to a FC SEMS, was excluded for analysis. In this patient the SEMS could not be inserted due to an acute cardiovascular event at the start of the endoscopic procedure. A total of 97 patients were included for final analysis, 48 patients in FC SEMS and 49 patients in the PC group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (11.4) | 69.2 (12.1) | 70.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 36 | 34 | 70
Dysphagia score [Mean (Standard Deviation); unit: units on a scale] — Dysphagia was scored according to the internationally used scoring system: score 0, able to consume a normal diet; score 1, dysphagia with certain solid foods; score 2, able to swallow semi-solid soft foods; score 3, able to swallow liquids only; score 4, complete dysphagia.
  Range 0-4, a higher score represents a worse outcome
  units on a scale | 2.8 (0.8) | 2.8 (0.7) | 2.8 (0.7)
WHO [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Performance Score
  0 Able to carry out all normal activity without restrictions.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out light work.
  2. Ambulatory and capable of all self-care but unable to carry out any work; up and more than 50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Range 0-4, a higher score respresents a worse outcome
  units on a scale | 1.4 (0.8) | 1.1 (0.8) | 1.3 (0.9)
Etiology/histology stricture [Count of Participants; unit: Participants]
  Adenocarcinoma | 24 | 32 | 56
  Squamous cell carcinoma | 22 | 13 | 35
  Extrinsic compression | 2 | 3 | 5
  Other | 1 | 0 | 1
Presence of distant metastasis [Number; unit: participants] | 30 | 30 | 60
Previous chemotherapy [Number; unit: participants] | 22 | 26 | 48
Previous radiotherapy [Number; unit: participants] | 19 | 18 | 37
Location stricture [Count of Participants; unit: Participants]
  Proximal esophagus | 7 | 8 | 15
  Mid esophagus | 12 | 13 | 25
  Distal esophagus or cardia | 30 | 27 | 57
Length of tumor [Mean (Standard Deviation); unit: cm] | 6.8 (3.1) | 7.6 (3.7) | 7.2 (3.5)
Length of stricture [Mean (Standard Deviation); unit: cm] | 5.4 (2.6) | 6.0 (2.9) | 5.7 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Dysphagia.
Description: This is defined as occurrence of dysphagia due to a stent or tumor related cause. These include tumor in- or overgrowth, stent migration, stent fracture or food impaction.
Time Frame: From stent placement (t=0) until death or placement of second stent, assessed up to 6 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS
Number analyzed (Participants) | 49 | 48
Participants | 11 | 9

2. Secondary Outcome: Number of Participants With Technical Success of SEMS Placement
Description: Technical succes was defined as succesful deployment of the stent which bridges the stricture
Time Frame: At stent placement (t=0)
Measure: Count of Participants; unit: Participants
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS
Number analyzed (Participants) | 49 | 48
Participants | 47 | 48

3. Secondary Outcome: Number of Participants With Clinical Success Defined as Improvement of Dysphagia Score
Description: Clinical success was defined as an improvement of dysphagia (at least 1 point reduction in the Dysphagia score) during follow-up.
  Dysphagia scores will be obtained at time point: t=0, t= 1 week, t=2 weeks, t=1 month, t=3 months and t= 6 months
Time Frame: From stent placement until death or placement of second stent, assessed up to 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS
Number analyzed (Participants) | 49 | 48
Participants | 43 | 40

4. Secondary Outcome: Number of Participants in Whom a Major Complication Has Occured
Description: A major adverse event was defined as a life-threatening event, including perforation, major haemorrhage, severe pain (NRS pain score ≥ 7), pneumonia, stridor and fistula.
Time Frame: From stent placement until death or placement of second stent, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS
Number analyzed (Participants) | 49 | 48
Participants | 23 | 18

5. Secondary Outcome: Median Survival After SEMS Placement
Description: Survival from stent placement until death or placement of second stent
Time Frame: From stent placement until death or placement of second stent
Measure: Median (Full Range); unit: days
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS
Number analyzed (Participants) | 49 | 48
days | 92 [5 to 656] | 61 [4 to 596]

ADVERSE EVENTS:
Description: One patient, which was allocated to a FC SEMS, was excluded for analysis. In this patient the SEMS could not be inserted due to an acute cardiovascular event at the start of the endoscopic procedure. A total of 97 patients were included for final analysis, 48 patients in FC SEMS and 49 patients in the PC group.
Arm/Group | Insertion of a Partially Covered SEMS | Insertion of a Fully Covered SEMS
Serious Adverse Events (participants affected / at risk) | 23/49 | 18/48
Other Adverse Events (participants affected / at risk) | 4/49 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insertion of a Partially Covered SEMS (N=49) | Insertion of a Fully Covered SEMS (N=48)
Severe pain (Gastrointestinal disorders) | 9 | 9
pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 | 4
mediastinitis (Gastrointestinal disorders) | 1 | 0
stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hemorrhage (Gastrointestinal disorders) | 5 | 4
Fistula (Gastrointestinal disorders) | 3 | 0
spondyloscitis (Musculoskeletal and connective tissue disorders) | 0 | 1
pressure ulcer (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insertion of a Partially Covered SEMS (N=49) | Insertion of a Fully Covered SEMS (N=48)
Fever (Infections and infestations) | 2 | 1
Mild pain (Gastrointestinal disorders) | 1 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes